CLINICAL TRIAL: NCT01487044
Title: A Single-Center Trial of High Frequency Pegaptanib for Rapid Restoration of VEGF Levels in Diabetic Retinal Edema
Acronym: GUARDIAN
Status: Available | Type: Expanded Access
Sponsor: Retina Institute of Hawaii (Other)
Collaborators: Eyetech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: RIH 1006
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Diabetic Macular Edema
Keywords: DME
MeSH Terms: interventions — pegaptanib

INTERVENTIONS:
Drug: Macugen (Pegaptanib Sodium) — Pegaptanib sodium drug substance is a pegylated (40 kDa branched PEG molecule consisting of two 20 kDa PEG arms) anti-VEGF aptamer. It is formulated in phosphate buffered saline at pH 6-7. Sodium hydroxide or hydrochloric acid may be added for pH adjustment.
  Pegaptanib sodium is formulated at 0.3mg/90µl and presented in USP Type I glass barrel syringes sealed with a bromobutyl rubber plunger stopper. The syringe has a needle attachment at allows for a 30-guage need to be fixed to the syringe prior to injection. The stoppered syringe is packaged in a foil pouch. The drug product is preservative-free and intended for single use by intravitreous injection only.

SUMMARY:
Establish the efficacy of initial high frequency loading of intravitreal pegaptanib bi-weekly during the initial treatment period when the VEGF levels are the greatest and then gradually extending the administration frequency to monthly as homeostasis ensues for the treatment of DME, as measured by best-corrected visual acuity.

DETAILED DESCRIPTION:
Determine if high frequency loading intravitreal pegaptanib will reduce the area and/or volume of DME, as assessed by Spectral Domain optical coherence tomography (SD-OCT) and to determine if this loading with gradual taper schedule of intravitreal pegaptanib will reduce the need for macular laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetics, with an age of 18 years of older
* Vision of 20/40-20/400 in the Study Eye
* Diabetic Macular Edema as documented by SD-OCT and Fluorescein Angiogram.

Exclusion Criteria:

* Cannot attened all trail required visits
* Eyes in which retinal surgery is needed now are is likely to be needed within 6 months, which the surgeon believes will not respond to non-surgical intervention.
* Presence of any abnormality that is likely to confound assessment of visual acuity improvement in eyes in which macular edema resolves, or improves, such as non-perfusion greater than 1 disc area involving the foveal avascular zone, epiretinal membrane associated with signs of contraction and/or significant opacification, or presence of chorioretinal atrophy involving the center of the macula.
* Vitreomacular traction determined clinically and/or by OCT, which, in the investigator's opinion, contributes to the macular edema, or causes associated foveal detachment, and would preclude improvement with pegaptanib sodium.
* Previous treatment with intravitreal corticosteroids in the study eye within 3 months of Day 0 visit.
* Previous treatment with intravitreal anti-angiogenic drugs in the study eye within 2 months of Day 0 visit.
* Previous intraocular surgery within 30 days of Day 0 visit.
* Any ocular or periocular infection within 30 days of Day 0 visit.
* Any of the following underlying diseases including:

History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 16.6), clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within 6 months, ventricular tachyarrythmias requiring ongoing treatment.

History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.

History or evidence of clinically significant impaired renal or hepatic function Stroke (within 12 months of trial entry). Any major surgical procedure within one month of trial entry.

* Any treatment with an investigational agent in the past 30 days for any condition.
* Known serious allergies to the fluorescein dye used in angiography or to the components of pegaptanib sodium formulation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Bennett, MD, Principal Investigator — Retina Institute of Hawaii
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States